CLINICAL TRIAL: NCT04533919
Title: Validation of Pre-Clinical Nano-Based Analgesics in Cells From Dorsal Root Ganglia
Brief Title: Validation of Pre-clinical Nano-Based Analgesics in Cells From Human Dorsal Root Ganglia
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0526; NCI-2020-05249 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0526 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-05; First posted 2020-09-01 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Neoplasm
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Dorsal root ganglia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Basic science (dorsal root ganglia collection): Patients' leftover dorsal root ganglia samples are collected during standard of care surgery.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of dorsal root ganglia

SUMMARY:
This study investigates the pre-clinical nano-based analgesics in cells from human dorsal root ganglia (clusters of neurons). Collecting these neurons may help future research related to safe and effective pain treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify translational mechanisms and therapeutics for neuropathic pain, a type of chronic pain that can arise due to injured nerves.

OUTLINE:

Patients' leftover dorsal root ganglia samples are collected during standard of care surgery.

ELIGIBILITY:
Inclusion Criteria:

---All patients undergoing surgery to resect spinal tumors

Exclusion Criteria:

---None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery to resect spinal tumors
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Viability assays | 3 years
  The Viability outcome measure will be expressed using percentage units. This will be calculated as the percentage of cells in culture that are able to exclude a cell permeable dye (Ethidium homodimer) from their nucleus. Entry of this dye into the nucleus and fluorescent binding to nuclear DNA is indicative of a dead/dying cell. Cultured cells that have undergone control or active nanoemulsion treatment in vitro will be loaded with a fluorescent calcium-sensitive dye and continuously monitored while excitation is evoked with a panel of ion channel agonists. The fold-change in intracellular calcium concentration over baseline in response to such excitation is the outcome measure.
Functional assays | 3 years
  Neurons will be isolated from fresh tissues and used in assays in which cells are stimulated with pronociceptive chemicals (e.g. agonists for ion channels, pattern recognition receptors, G protein-coupled receptors). Cell activity will be quantified as appropriate (e.g. calcium mobilization). Experimental endpoints will be analyzed using a between-subjects designs to assess differences between patients with and without nerve compression. ANOVA will be performed in a 2 (neuropathic pain vs. control) x 4 (3 treatments vs. control) design. Bonferroni posthoc tests will be applied when significant interactions are found. Age, sex, ethnicity, cancer diagnosis, drug treatments, and history of chronic pain will be included as covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Shepherd, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: http://www.mdanderson.org — http://www.mdanderson.org